CLINICAL TRIAL: NCT03007550
Title: Prospective Randomized Controlled Multicenter Clinical Trial For Comparison Of Safety Between Laparoscopic And Open Total Gastrectomy In Patients With Clinical Stage I Gastric Cancer
Brief Title: Study On Safety Of Laparoscopic Total Gastrectomy For Clinical Stage I Gastric Cancer
Acronym: CLASS02-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Yihong Sun, Clinical Professor,Department of General Surgery, Zhongshan Hospital, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZSGC-001
Record Dates: First submitted 2016-12-22; First posted 2017-01-02 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Laparoscopic total gastrectomy; Open total gastrectomy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic total gastrectomy (Experimental): The surgeon will perform LTG with D1+/D2-10 lymphadenectomy for patients enrolled in this group.
  Interventions: Procedure: Laparoscopic total gastrectomy
- Open total gastrectomy (Other): The surgeon will perform OTG with D1+/D2-10 lymphadenectomy for patients enrolled in this group.
  Interventions: Procedure: Open total gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic total gastrectomy — LTG with D1+/D2-10 lymphadenectomy for patients with clinical stage I (T1N0M0、T1N1M0、T2N0M0) gastric adenocarcinoma
  Other Names: Study group (LTG)
  Arms: Laparoscopic total gastrectomy
Procedure: Open total gastrectomy — OTG with D1+/D2-10 lymphadenectomy for patients with clinical stage I (T1N0M0、T1N1M0、T2N0M0) gastric adenocarcinoma
  Other Names: Control group (OTG)
  Arms: Open total gastrectomy

SUMMARY:
This CLASS02-01 trial is a prospective, multicenter trial for laparoscopic total gastrectomy (LTG) and open total gastrectomy (OTG) in patients with clinical stage I (T1N0M0、T1N1M0、T2N0M0) gastric cancer. The primary purpose of this study is to evaluate the early operative morbidity and mortality and determine the safety of LTG compared with OTG for clinical stage I gastric adenocarcinoma. The second purpose is to evaluate the recovery course and compare the postoperative hospital stay of the patients enrolled in this study.

DETAILED DESCRIPTION:
Gastric cancer is an important health problem, being the fourth most common cancer and the third leading cause of cancer-related death worldwide. Age standardized mortality rates for gastric cancer are 14.3 per 100 000 in men and 6.9 per 100 000 in women. Incidence shows clear regional and sex variations-rates are highest in Eastern Asia, Eastern Europe, and South America and lowest in Northern and Southern Africa. More than 679 000 new cases and 498,000 deaths occur every year in China, and an increasing trend of proximal gastric cancer is observed during the past years.

More than 20 years after the introduction of laparoscopic gastrectomy, many large-scale randomized controlled trials have been conducted in Japan (JCOG0912 and JLSSG0901), Korea (KLASS01 and KLASS02), and China (CLASS01). These trials are all designed to evaluate the non-inferiority of laparoscopic-assisted distal gastrectomy (LADG) to its open counterpart. No RCT for laparoscopic total gastrectomy (LTG) exists at this moment. The standardization of techniques for esophagojejunal anastomosis in LTG has been difficult even for experienced surgeons.

At present, Japan (JCOG1401), Korea (KLASS03), and Netherlands (STOMACH) have planned or launched clinical studies on LTG. China is one of the countries with the highest incidence of gastric cancer and surgeons have accumulated extensive experience through CLASS01 study. So, it's time for conducting the clinical research on the safety of LTG for gastric cancer.

This CLASS02-01 trial is a prospective, multicenter trial for LTG and open total gastrectomy (OTG) in patients with clinical stage I (T1N0M0、T1N1M0、T2N0M0) gastric cancer. The primary purpose of this study is to evaluate the early operative morbidity and mortality and determine the safety of LTG compared with OTG for clinical stage I gastric adenocarcinoma. The second purpose is to evaluate the recovery course and compare the postoperative hospital stay of the patients enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years；
2. Primary lesion is pathologically diagnosed as gastric adenocarcinoma, such as papillary adenocarcinoma, tubular adenocarcinoma, mucinous adenocarcinoma, poorly cohesive carcinoma (including signet ring cell carcinoma and other variants), and mixed adenocarcinoma;
3. Clinical stage IA (T1N0M0) or IB (T1N1M0, T2N0M0) (According to AJCC-7th TNM staging system);
4. Tumor located in the upper or middle third of the stomach, and curative resection is expected to be achievable by total gastrectomy with D1+/D2-10 lymphadenectomy (also apply to multiple primary cancers);
5. No invasion to Z-line;
6. BMI (Body Mass Index) < 30 kg/m2;
7. No history of upper abdominal surgery (except for laparoscopic cholecystectomy);
8. No prior treatment of chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc.;
9. No enlargement of splenic hilar lymph nodes;
10. Preoperative performance status (ECOG，Eastern Cooperative Oncology Group) of 0 or 1;
11. Preoperative ASA (American Society of Anesthesiologists) scoring: I-III;
12. Sufficient organ functions;
13. Written informed consent.

Exclusion Criteria:

1. Preoperative examinations indicate that the stage of the disease is stage II/III/IV;
2. Preoperative examination indicate enlargement of perigastric or retroperitoneal lymph nodes (min diameter≥1.0cm);
3. Women during pregnancy or breast-feeding;
4. Synchronous or metachronous (within 5 years) malignancies;
5. Body temperature ≥ 38℃ before surgery or infectious disease with a systemic therapy indicated;
6. Severe mental disease;
7. Severe respiratory disease;
8. Severe hepatic and renal dysfunction;
9. Unstable angina pectoris or history of myocardial infarction within 6 months;
10. History of cerebral infarction or cerebral hemorrhage within 6 months;
11. Continuous systemic steroid therapy within 1 month (except for topical use);
12. Gastric cancer complications (bleeding, perforation, obstruction) that requiring emergency surgery;
13. Patients are participating or have participated in another clinical trial (within 6 months).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Early operative morbidity and mortality rate | 30 days
  The early operative morbidity and mortality are defined as the event observed within 30 days following surgery, including intraoperative and postoperative complications and/or death.

SECONDARY OUTCOMES:
Postoperative recovery course | 30 days
  Time to first ambulation, flatus, liquid diet, and soft diet are used to assess the postoperative recovery course, which is a composite outcome measure.
Postoperative hospital stay | 30 days
  The length of postoperative hospital stay will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Yihong Sun, MD, Principal Investigator — Fudan University
Locations (1):
- ZhongShan hospital FuDan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Kim HH, Hyung WJ, Cho GS, Kim MC, Han SU, Kim W, Ryu SW, Lee HJ, Song KY. Morbidity and mortality of laparoscopic gastrectomy versus open gastrectomy for gastric cancer: an interim report--a phase III multicenter, prospective, randomized Trial (KLASS Trial). Ann Surg. 2010 Mar;251(3):417-20. doi: 10.1097/SLA.0b013e3181cc8f6b. PMID 20160637
- [Background] Chen K, Xu XW, Zhang RC, Pan Y, Wu D, Mou YP. Systematic review and meta-analysis of laparoscopy-assisted and open total gastrectomy for gastric cancer. World J Gastroenterol. 2013 Aug 28;19(32):5365-76. doi: 10.3748/wjg.v19.i32.5365. PMID 23983442
- [Background] Kim HH, Han SU, Kim MC, Hyung WJ, Kim W, Lee HJ, Ryu SW, Cho GS, Kim CY, Yang HK, Park DJ, Song KY, Lee SI, Ryu SY, Lee JH; Korean Laparoscopic Gastrointestinal Surgery Study (KLASS) Group. Prospective randomized controlled trial (phase III) to comparing laparoscopic distal gastrectomy with open distal gastrectomy for gastric adenocarcinoma (KLASS 01). J Korean Surg Soc. 2013 Feb;84(2):123-30. doi: 10.4174/jkss.2013.84.2.123. Epub 2013 Jan 29. PMID 23396494
- [Background] Nakamura K, Katai H, Mizusawa J, Yoshikawa T, Ando M, Terashima M, Ito S, Takagi M, Takagane A, Ninomiya M, Fukushima N, Sasako M. A phase III study of laparoscopy-assisted versus open distal gastrectomy with nodal dissection for clinical stage IA/IB gastric Cancer (JCOG0912). Jpn J Clin Oncol. 2013 Mar;43(3):324-7. doi: 10.1093/jjco/hys220. Epub 2012 Dec 28. PMID 23275644
- [Background] Jeong O, Ryu SY, Choi WY, Piao Z, Park YK. Risk factors and learning curve associated with postoperative morbidity of laparoscopic total gastrectomy for gastric carcinoma. Ann Surg Oncol. 2014 Sep;21(9):2994-3001. doi: 10.1245/s10434-014-3666-x. Epub 2014 Apr 1. PMID 24687152
- [Background] Kim HH, Han SU, Kim MC, Hyung WJ, Kim W, Lee HJ, Ryu SW, Cho GS, Song KY, Ryu SY. Long-term results of laparoscopic gastrectomy for gastric cancer: a large-scale case-control and case-matched Korean multicenter study. J Clin Oncol. 2014 Mar 1;32(7):627-33. doi: 10.1200/JCO.2013.48.8551. Epub 2014 Jan 27. PMID 24470012
- [Background] Kim HI, Hur H, Kim YN, Lee HJ, Kim MC, Han SU, Hyung WJ. Standardization of D2 lymphadenectomy and surgical quality control (KLASS-02-QC): a prospective, observational, multicenter study [NCT01283893]. BMC Cancer. 2014 Mar 19;14:209. doi: 10.1186/1471-2407-14-209. PMID 24646327
- [Background] Villanueva MT. Gastric cancer: a master KLASS in laparoscopic gastrectomy. Nat Rev Clin Oncol. 2014 Mar;11(3):119. doi: 10.1038/nrclinonc.2014.18. Epub 2014 Feb 11. No abstract available. PMID 24514147
- [Background] Wada N, Kurokawa Y, Takiguchi S, Takahashi T, Yamasaki M, Miyata H, Nakajima K, Mori M, Doki Y. Feasibility of laparoscopy-assisted total gastrectomy in patients with clinical stage I gastric cancer. Gastric Cancer. 2014 Jan;17(1):137-40. doi: 10.1007/s10120-013-0235-0. Epub 2013 Feb 22. PMID 23430265
- [Background] Byun C, Han SU. Current status of randomized controlled trials for laparoscopic gastric surgery for gastric cancer in Korea. Asian J Endosc Surg. 2015 May;8(2):130-8. doi: 10.1111/ases.12176. Epub 2015 Mar 5. PMID 25753372
- [Background] Hur H, Lee HY, Lee HJ, Kim MC, Hyung WJ, Park YK, Kim W, Han SU. Efficacy of laparoscopic subtotal gastrectomy with D2 lymphadenectomy for locally advanced gastric cancer: the protocol of the KLASS-02 multicenter randomized controlled clinical trial. BMC Cancer. 2015 May 5;15:355. doi: 10.1186/s12885-015-1365-z. PMID 25939684
- [Background] Inaki N, Etoh T, Ohyama T, Uchiyama K, Katada N, Koeda K, Yoshida K, Takagane A, Kojima K, Sakuramoto S, Shiraishi N, Kitano S. A Multi-institutional, Prospective, Phase II Feasibility Study of Laparoscopy-Assisted Distal Gastrectomy with D2 Lymph Node Dissection for Locally Advanced Gastric Cancer (JLSSG0901). World J Surg. 2015 Nov;39(11):2734-41. doi: 10.1007/s00268-015-3160-z. PMID 26170158
- [Background] Katai H. Current status of a randomized controlled trial examining laparoscopic gastrectomy for gastric cancer in Japan. Asian J Endosc Surg. 2015 May;8(2):125-9. doi: 10.1111/ases.12171. Epub 2015 Feb 10. PMID 25676458
- [Background] Lee JH, Nam BH, Ryu KW, Ryu SY, Park YK, Kim S, Kim YW. Comparison of outcomes after laparoscopy-assisted and open total gastrectomy for early gastric cancer. Br J Surg. 2015 Nov;102(12):1500-5. doi: 10.1002/bjs.9902. Epub 2015 Sep 23. PMID 26398912
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Hu Y, Huang C, Sun Y, Su X, Cao H, Hu J, Xue Y, Suo J, Tao K, He X, Wei H, Ying M, Hu W, Du X, Chen P, Liu H, Zheng C, Liu F, Yu J, Li Z, Zhao G, Chen X, Wang K, Li P, Xing J, Li G. Morbidity and Mortality of Laparoscopic Versus Open D2 Distal Gastrectomy for Advanced Gastric Cancer: A Randomized Controlled Trial. J Clin Oncol. 2016 Apr 20;34(12):1350-7. doi: 10.1200/JCO.2015.63.7215. Epub 2016 Feb 22. PMID 26903580
- [Background] Jung DH, Son SY, Park YS, Shin DJ, Ahn HS, Ahn SH, Park DJ, Kim HH. The learning curve associated with laparoscopic total gastrectomy. Gastric Cancer. 2016 Jan;19(1):264-72. doi: 10.1007/s10120-014-0447-y. Epub 2014 Dec 7. PMID 25481705
- [Background] Kim W, Kim HH, Han SU, Kim MC, Hyung WJ, Ryu SW, Cho GS, Kim CY, Yang HK, Park DJ, Song KY, Lee SI, Ryu SY, Lee JH, Lee HJ; Korean Laparo-endoscopic Gastrointestinal Surgery Study (KLASS) Group. Decreased Morbidity of Laparoscopic Distal Gastrectomy Compared With Open Distal Gastrectomy for Stage I Gastric Cancer: Short-term Outcomes From a Multicenter Randomized Controlled Trial (KLASS-01). Ann Surg. 2016 Jan;263(1):28-35. doi: 10.1097/SLA.0000000000001346. PMID 26352529
- [Background] Huang CM, Zhang JR, Zheng CH, Li P, Xie JW, Wang JB, Lin JX, Lu J, Chen QY. A 346 case analysis for laparoscopic spleen-preserving no.10 lymph node dissection for proximal gastric cancer: a single center study. PLoS One. 2014 Sep 29;9(9):e108480. doi: 10.1371/journal.pone.0108480. eCollection 2014. PMID 25264673
- [Background] Kurokawa Y, Katai H, Fukuda H, Sasako M; Gastric Cancer Surgical Study Group of the Japan Clinical Oncology Group. Phase II study of laparoscopy-assisted distal gastrectomy with nodal dissection for clinical stage I gastric cancer: Japan Clinical Oncology Group Study JCOG0703. Jpn J Clin Oncol. 2008 Jul;38(7):501-3. doi: 10.1093/jjco/hyn055. Epub 2008 Jun 26. PMID 18586666
- [Derived] Liu F, Huang C, Xu Z, Su X, Zhao G, Ye J, Du X, Huang H, Hu J, Li G, Yu P, Li Y, Suo J, Zhao N, Zhang W, Li H, He H, Sun Y; Chinese Laparoscopic Gastrointestinal Surgery Study (CLASS) Group. Morbidity and Mortality of Laparoscopic vs Open Total Gastrectomy for Clinical Stage I Gastric Cancer: The CLASS02 Multicenter Randomized Clinical Trial. JAMA Oncol. 2020 Oct 1;6(10):1590-1597. doi: 10.1001/jamaoncol.2020.3152. PMID 32815991
- [Derived] He H, Li H, Su X, Li Z, Yu P, Huang H, Huang C, Ye J, Li Y, Suo J, Yu J, Li G, Xu Z, Zhao G, Cao H, Hu J, Du X, Liu F, Sun Y; Chinese Laparoscopic Gastrointestinal Surgery Study (CLASS) Group. Study on safety of laparoscopic total gastrectomy for clinical stage I gastric cancer: the protocol of the CLASS02-01 multicenter randomized controlled clinical trial. BMC Cancer. 2018 Oct 3;18(1):944. doi: 10.1186/s12885-018-4846-z. PMID 30285673